CLINICAL TRIAL: NCT03128294
Title: Long Term Survivors in Ovarian Cancer
Status: Terminated | Type: Observational
Why Stopped: Data was not sufficiently complete and reliable for analysis (retrospective chart research)
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201600799
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- long-term survivors of ovarian cancer: long-term survivors of ovarian cancer
  Interventions: Other: Retrospective, cross-sectional descriptive analysis

INTERVENTIONS:
Other: Retrospective, cross-sectional descriptive analysis — This study is a retrospective, cross-sectional descriptive analysis, and concerns the extraction of data from anonymised patient files. A database will be constructed and descriptive statistics will be used to summarise the data.

SUMMARY:
In this study the investigators would like to explore the patient and tumour characteristics of long-term survivors of ovarian cancer (>10 years). Indentifiying the characteristics of long-term survivors not only helps find prognostic factors for survival but may aid in generating hypotheses for novel therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

To achieve a large enough study population of approximately 80 subjects, patients surviving >10 years after treatment for stage IIIC/IV epithelial ovarian cancer in the past 25 years will be included from five hospitals. Patients were diagnosed between 1979 and 2006 and treated in the north of the Netherlands. A list of subjects fitting these inclusion criteria will be extracted from the National Cancer Registry (NKR).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Long-term survivors of ovarian cancer (>10 years).
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Indentifiying the characteristics of long-term survivors | 2 years
  Indentifiying the characteristics of long-term survivors

CONTACTS AND LOCATIONS:
Overall Officials: A.K.L. Reyners, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands